CLINICAL TRIAL: NCT02086487
Title: Efficacy and Safety Assessment of NIlotinib in CML Patients With Suboptimal Response on Imatinib Therapy (NISRI)
Brief Title: Efficacy and Safety Assessment of NIlotinib in CML Patients With Suboptimal Response on Imatinib Therapy
Acronym: NISRI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of many unseen obstacles resulted in poor accrual, study is terminated.
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC12/052
Record Dates: First submitted 2014-02-27; First posted 2014-03-13 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: NIlotinib , Suboptimal Response , Imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib 300 mg (Experimental): Patients diagnosed with chronic myeloid leukemia receiving treatment of Imatinib 400 mg but show sub-optimal response on Imatinib therapy as per the ELN 2013 guidelines will be switched to Nilotinib 300 mg twice daily and will be assessed for timely.
  In the absence of safety concerns, nilotinib could be escalated to 400 mg twice daily if patients had not obtained any of the following milestones:
  1. BCR-ABL1 transcript level ≤ 10% at 3 months;
  2. CCyR at 6 months,
  3. BCR/ABL1 ≤ 1% at 6 months
  4. MMR at 12 months, or
  5. if they showed loss of cytogenetic or molecular response or disease progression at any time. Failure and thus, stopping nilotinib will be considered if any of above milestones happened while on the 400mg twice daily dose.
  Interventions: Drug: Nilotinib 300 mg.

INTERVENTIONS:
Drug: Nilotinib 300 mg. — Patients diagnosed with chronic myeloid leukemia receiving treatment of Imatinib 400 mg once a day but are determined to be sub-optimally responding to Imatinib therapy as per the ELN 2013 guidelines will be switched to Nilotinib 300 mg BID and then will be assessed for therapy response. ELN guidelines 2013 for imatinib therapy response states as:
  Minor cytogenetic response mCyR or minimal response at 3 months (Ph+ metaphases in BM 35 to 95 %); BCR-ABL1 transcript > 10% at 3 months; Partial cytogenetic response at 6 months Ph+ metaphases in BM 0to 35); BCR-ABL1 transcript is 1 to 10% at 6 months. Less than a major molecular response at > 12 months; i.e (BCR-ABL1 0.1 -1%)
  Other Names: Tasigna 300 mg

SUMMARY:
whether Nilotinib at the two sequential dosage forms will induce quicker and deeper response in those patients, and if FISH on PB (Peripheral blood) would be an effective way to monitor response compared to conventional cytogenetics on bone marrow (BM) sample

DETAILED DESCRIPTION:
This is a multicenter, open label trial which will be conducted within Kingdom of saudi Arabia for which CML (Chronic Myeloid Leukemia) patients who meet eligibility criteria and showing sub optimal response to Imatinib therapy as per European leukemia Net ELN 2013 guidelines will be recruited and switched to Nilotinib 300 mg twice a day therapy.

Efficacy assessments of hematologic and cytogenetic response and disease progression, will be performed every 6 months at a minimum, including hematologic analysis, bone marrow cytogenetics, and molecular studies to ensure that nilotinib is being provided to patients who were responding and that patients who progressed could discontinue therapy.

Safety assessments include evaluation of adverse events, hematologic assessment, biochemical testing, cardiac enzyme assessment, serial electrocardiogram evaluation, and physical examination. Adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0. Survival will be dated from start of nilotinib therapy until death from any cause and censored at last follow-up for patients who were alive.

The data will be summarized with respect to demographic and baseline characteristics, efficacy evaluation, and safety observations and measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study procedures being performed.
2. Age 18 or above of male or female CML patients in chronic phase.
3. Eastern Cooperative Oncology Group ECOG Performance status 0, 1 or 2
4. Sub-optimal response on Imatinib therapy as determined by any of the following criteria: 4.1) Minor cytogenetic response mCyR or minimal response at 3 months (Ph+ metaphases in BM 35 to 95 %) 4.2) BCR-ABL1 transcript >10% at 3 months; 4.3) Partial cytogenetic response PCyR at 6 months; (i.e Ph+ metaphases in BM 0 to 35%) 4.4) BCR-ABL1 transcript 1 - 10% at 6 months 4.5) Less than a major molecular response at > 12 months; i.e (BCR-ABL1 0.1 - 1%)
5. Normal serum levels of potassium, magnesium and calcium ≥ LLN (lower limit of normal) or corrected to within normal limits with supplements, prior to the first dose of study medication,
6. Aspartate aminotransferase AST and Alanine aminotransferase ALT ≤ 2.5 x ULN (upper limit of normal)
7. Alkaline phosphatase ≥ 2.5 x ULN
8. Total bilirubin ≤ 1.5 x ULN;
9. Serum amylase ≤ 1.5 x ULN Performance status ECOG 0,1,2

Exclusion Criteria:

1. Previous Exposure to Tyrosine Kinase Inhibitor (TKI) other than Imatinib for more than 2 weeks
2. Patients who are already participating in any other clinical trial.Patients who were not compliant to Imatinib therapy.
3. Optimal response to Imatinib therapy as determined by any one of the criteria: 3.1. CCyR or PCyR at 3 months (Ph+ metaphases in BM ≤ 35 %). 3.2. BCR-ABL1 transcript ≤ 10 % at 3 months. 3.3. CCyR at 6 months (Ph+ metaphases in BM 0 %). 3.4. BCR-ABL1 transcript < 1% at 6 months. 3.5. BCR-ABL1 transcript ≤ 0.1 % at 12 months. 3.6. BCR-ABL1 transcript ≤ 0.1 % at any time.
4. Failure response to Imatinib therapy as per ELN guidelines 2013 as determined by any of the criteria: 4.1. Non- complete hematologic response (Non- CHR) or no cytogenetic response CyR at 3 months (Ph+ metaphases in BM > 95 %). 4.2. Less than Partial cytogenetic response PCyR at 6 months (Ph+ metaphases in BM > 35%). 4.3. BCR-ABL1 transcript >10 % at 6 months. 4.4. Less than complete cytogenetic response CCyR at 12 months (Ph+ metaphases in BM > 0 %). 4.5. BCR-ABL1 transcript >1 % at 12 months. 4.6. Loss of CHR or loss of CCyR or confirmed loss of MMR* or development of partially imatinib - sensitive BCR-ABL mutation or CCA in Ph- positive cells at any time.
5. Pregnant or lactating females
6. Patients with prolonged QT intervals
7. Patient with history of pancreatitis
8. Previously documented T315I mutations;
9. Uncontrolled congestive heart failure or hypertension;
10. Myocardial infarction or unstable angina pectoris within past 12 months;
11. Significant arrhythmias, including history or presence of clinically significant ventricular or atrial tachyarrhythmias, clinically -significant bradycardias, long QT syndrome and/or corrected QT interval (QTc) > 450 msec on screening ECG. Patients with complete LBBB (Left Bundle Branch Block);
12. Patients concurrently on strong CYP3A4 inhibitors.
13. Other concurrent uncontrolled medical conditions (e.g. uncontrolled diabetes, active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol;
14. Impaired gastrointestinal function or GI disease that may alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric by-pass surgery);
15. Patients with another primary malignancy that is currently clinically significant or requires active intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable of this study is the overall Major molecular response at 12 month after starting Nilotinib 300mg twice daily for patient who suboptimally responded to Imatinib as per the ELN guidelines | 12 Months

SECONDARY OUTCOMES:
Rate of cytogenetic response (complete cytogenetic response CCyR and Major cytogenetic response MCyR) and Major molecular response MMR at 3, 6 and 12 months of starting Nilotinib in patients who had a suboptimal response on Imatinib. | 12Months
Rate of CCyR at 6 months and MMR at 6 and 12 months from Nilotinib dose escalating to 400 mg BID. | 12 months
Rate and duration of Complete Hematologic Response CHR. | 12 months
Rate of CMR at 12 months of Nilotinib. | 12 months
Comparison of FISH results with conventional cytogenetics at 3, 6 & 12 months. | 12
Overall survival. | 12

OTHER OUTCOMES:
Mutational analysis for the patients with suboptimal response at the pre defined end points as per the ELN guidelines. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ahmad S. Alaskar, MD,FACP,FRCP, Principal Investigator — King Abdulaziz Medical City
Locations (2):
- Saudi Arabia (2):
  - National Guard Hospital, Riyadh, Central
  - King Fahad specialist Hospital, Dammam, Eastern Province

IPD SHARING:
Plan to Share IPD: Undecided